CLINICAL TRIAL: NCT06746350
Title: Feasibility of Integrating Thermotherapy (TT) for Treatment of Cutaneous Leishmaniasis Into the Primary Healthcare Facilities in East Gurage Zone, Ethiopia
Brief Title: Feasibility of Integrating Thermotherapy for Treatment of Cutaneous Leishmaniasis in Primary Health Care Setup
Acronym: TTCL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Armauer Hansen Research Institute, Ethiopia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TTCL; TTCL (Other: AHRI)
Record Dates: First submitted 2024-12-04; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Cutaneous Leishmaniasis; Sodo; Thermotherapy; ThermoMed
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Hyperthermia | interventions — Hyperthermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thermotherapy (Experimental): This arm receives thermotherapy right after CL diagnosis
  Interventions: Device: Thermotherapy
- Control group for three months (Other): This arm receives thermotherapy three-month after CL diagnosis.
  Interventions: Device: Thermotherapy

INTERVENTIONS:
Device: Thermotherapy — Radio frequency-induced heat treatment using the ThermoMed device at 50-degree centigrade for 30 seconds.
  Other Names: ThermoMed™

SUMMARY:
This study will look at how practical it is to use thermotherapy (TT) as a treatment for skin(cutaneous) leishmaniasis (CL) in health centers in the Sodo and South Sodo districts, Ethiopia. The main questions the investigators want to answer are:

* Is it practical, acceptable, and suitable to use thermotherapy for treating skin leishmaniasis in these health centers?
* How effective is thermotherapy in treating skin leishmaniasis in this setting?

Health centers that do not offer thermotherapy will be used as a comparison group. Patients with CL in these areas will be monitored for up to 3 months before being sent to centers that provide thermotherapy.

Participants will be checked at a nearby health center to see if they meet the criteria for the study and then recruited. Patients with skin lesions will receive thermotherapy using the ThermoMed device, which heats the area to 50°C for 30 seconds. Their progress will be checked every 4 weeks until day 90. Depending on how well they respond, thermotherapy may be repeated at 4 or 8 weeks.

DETAILED DESCRIPTION:
This study aims to improve access to effective treatment for cutaneous leishmaniasis (CL), specifically focusing on treatment with thermotherapy (TT) in selected districts in Sodo and south Sodo districts in Ethiopia. The study is structured into three phases, aligned with the different phases of the MRC framework for complex interventions. It follows an iterative approach, where the following phases depend on the findings from the preceding phases.

* Phase 1 of the project works on developing the training packages for the PHC staff and Health Extension Workers (HEWs) to diagnose/manage patients with CL and to refer suspected CL patients to the health centers respectively. The investigators will develop the training packages in consultation with a dermatologist with experience in TT for CL, the research team, the health department officials, the primary healthcare (PHC) staff, and HEWs.
* Phase 2- involves piloting the intervention approach in two of the health centers and TT will be administered by the PHC staff for 20 CL patients. In this phase, the investigators will do a feasibility, acceptability, and appropriateness assessment. The feasibility assessments encompass technical and allocative. Technical feasibility assesses the match between the technical complexity of the intervention and the capacity to implement it while allocative feasibility assesses whether the right approach is being followed in terms of resource allocation within the healthcare system. The PHC staff who have experience implementing TT and the health officials will be in a better position to give this critical information in a focus group discussion. The investigators will also assess fidelity to assess whether the training package has been well received by the PHC staff.

Phase 3- involves implementing the intervention in other health centers and on larger CL patients and assessing the feasibility, acceptability, appropriateness, as well as cost-effectiveness. In this phase, TT treatment will be administered to an additional 145 people making the total number of CL patients treated in this study 165. While implementing the study activities, we will abide by the Good Clinical Practice (GCP) principles. Serious and Unexpected Serious Adverse Reactions (SUSARs) will also be reported to the Ethiopian Food and Drug Authority (EFDA) according to the pharmacovigilance requirement of the Authority.

In this study, the following research designs will be followed:

1. Qualitative study designs; The researchers will use Focus Group Discussions (FGDs) to assess the feasibility, acceptability, and appropriateness of integrating TT from the PHC staff, the health officials, and HEWs. Additionally, to assess the same parameters from patients and the community in-depth interviews will employed. To further augment data collected through FGD and in-depth interviews to assess feasibility, acceptability, and appropriateness using a validated tool by Weiner et al. The investigators will assess fidelity to evaluate to what extent the trained PHC staff has adhered to the training package which could also tell us the technical feasibility of the intervention. The feasibility assessment includes allocative and technical feasibility.
2. A cross-sectional study to assess the diagnostic accuracy of primary health care staff in correctly identifying CL patients using PCR as a gold standard. This design will assist in further assessing the fidelity of the PHC staff in adhering to the training package delivered in the first phase of the training. Additionally, the investigators will have information on the technical feasibility of the intervention by looking at the percentage of CL cases and non-CL cases correctly identified.
3. Quasi-experimental design to assess the treatment success rate of TT in treating CL. An independent dermatologist will assess the response to the TT. In this study, there is neither a control group nor randomized patients The catchment areas of health centers that are not providing TT will serve as a control group. Patients with CL within these control catchment areas will be followed for a maximum of 3 months before they are referred to TT-providing centers for treatment. Eligible CL patients are offered TT treatment by the PHC staff and only if interested, the CL Patients will undergo TT treatment. TT will be administered up to two times to the Cutaneous Leishmaniasis (CL) patients in the intervention group:

   * CL patients who do not show a response during their week 4 visit will receive a second dose of TT at the same visit.
   * CL patients who show an initial response at week 4, will be assessed further during their week 8 visit. If it is unlikely that the patients will achieve complete epithelialization of their ulcers or flattening of their nodules within the next 4 weeks, they will receive a second dose of TT during that same week 8 visit.

   Patients will be followed for response to treatment. In addition to allowing the targets for the qualitative studies to experience first-hand the effects of TT, this part of the study further helps in indirectly verifying whether the PHC staff are adhering to the training on the administration of TT and the technical feasibility of TT administration.
4. A cross-sectional study to assess the diagnostic accuracy of AI-based CL diagnosis using PCR as a gold standard. If this approach is proven to work, then deployment of thermotherapy in the study area will be further facilitated without a need for laboratory confirmation of CL.

PHC staff, i.e. general practitioners, health officers, and/or nurses, will be trained on the spot diagnosis of CL, taking digital pictures of lesions, taking scrape samples from the lesions, as well as administration of TT to the suspected CL lesions with the training package developed under phase 1 of the study. Then the primary healthcare staff, as per their training, will make clinical suspicion of CL and apply TT on the suspected CL lesions. Suspected CL lesions will also be followed for up to a maximum of 180 days. Before administering TT, the primary healthcare staff will take good-quality digital pictures and skin scrape samples from the suspected CL lesions for later confirmation with PCR. HEWs, who are based in the health posts, will be an integral part of the whole process by sending possible cases of CL to the primary healthcare facilities for initial diagnosis as well as sensitizing the patients for follow up visits. The investigators will carefully choose two to three primary health care facilities located in areas with a notably higher occurrence of CL within their catchment areas for the implementation of CL diagnosis and TT application. The deployment of ThermoMed™ devices will initially occur at these selected facilities. CL patients living within the catchment areas of the remaining health centers that are not providing the TT intervention will serve as the control group. These control group patients will be observed for a maximum of three months and they will be referred to TT-providing centers for treatment. Patients in the control group have the right to seek CL treatment on their own during this observation period. If the flow of CL patients at these facilities is considered insufficient, there is a possibility of relocating the ThermoMed™ devices to other primary healthcare facilities in Sodo and South Sodo. An equal number of digital pictures of and scrape samples from the lesions of participants suspected to have skin diseases other than CL will be collected for comparison. TT will be administered using a radio frequency-induced heat therapy (RFHT) by a ThermoMed™ device (Thermosurgery Technologies, Inc., Phoenix, AZ). RFHT is applied only once for 30 seconds at 500C. TT could also be delivered by handheld exothermic crystallization thermotherapy for CL (HECT-CL) device. However, since HECT-CL needs repeated applications up to seven times and due to its lower rate of efficacy compared to RHFT, the researchers decided to use ThermoMed™. Patients who are successfully treated with TT will be visited on day 180 to see if the lesions relapse.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged ≥12 and ≤60 years old.
* Patient has a lesion that satisfies the following criteria:

  * Lesion size < or = 4 cm (longest diameter).
  * Not located adjacent to ear, nose, eyes, lips, or close to mucosal membranes.
  * Patient with < or = 4 CL lesions
* Patient able to give written informed consent.

Exclusion Criteria:

* Any condition that prevents the patient from following the study treatment and/or the follow-up

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2026-05-25 (Estimated); Study Completion 2027-05-25 (Estimated)

PRIMARY OUTCOMES:
Feasibility, acceptability, and appropriateness of integrating TT into primary healthcare. | Day 90 reached for 20 patients
  - Focus Group Discussion (FGD) and in-depth interview
Feasibility, acceptability, and appropriateness of integrating TT into primary healthcare. | Day 90 reached for 20 patients
  Assessment of Feasibility of Intervention Measure (FIM), Acceptability of Intervention Measure (AIM), and Intervention Appropriateness Measure (IAM) using a validated psychometric tool.

SECONDARY OUTCOMES:
Treatment success rate | Day 90 reached for all patients
  The proportion of patients who are cured at day 90. Cure is defined as complete epithelialization for ulcer lesions and complete flattening of nodules.
Diagnostic accuracy of primary health care staff | Day 0 for all the participants reached
  Calculating sensitivity, specificity, positive, and negative predictive values of CL diagnosis by primary healthcare staff using PCR as a gold standard.
Diagnostic accuracy of AI in making a diagnosis of CL | Day 0 for all the participants reached
  Calculating sensitivity, specificity, positive, and negative predictive values of CL diagnosis by AI-based program using PCR as a gold standard.

IPD SHARING:
Plan to Share IPD: Undecided
We don't have a plan to share IPD at the current moment.